CLINICAL TRIAL: NCT03111095
Title: Remote Patient Monitoring - Telehealth for Management of Women With Postpartum Hypertension
Brief Title: Postpartum Hypertension: Remote Patient Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-003
Record Dates: First submitted 2017-03-24; First posted 2017-04-12 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-07

CONDITIONS: Hypertension, Pregnancy-Induced
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Participants (Experimental): Subjects will use the mobile health device to record their blood pressure and weight measurements everyday for 6 weeks postpartum.
  Interventions: Other: Mobile Health
- Standard of Care (No Intervention): This arm is a chart review done on hypertensive women who do not participate in using the mobile health device.

INTERVENTIONS:
Other: Mobile Health — Subjects will submit blood pressure and weight measurements daily for 6 weeks postpartum. Subjects will have a video telehealth visit with the mobile health nurse at 48 hours and 7 days after discharge from the hospital.
  Arms: Mobile Health Participants

SUMMARY:
The purpose of this study is to see if Honeywell Genesis Android Touch Bluetooth System (mobile health) can improve patient satisfaction and quality of care provided to women experiencing complications due to high blood pressure during pregnancy.

DETAILED DESCRIPTION:
For six weeks postpartum, patients will use Honeywell Genesis Android Touch Bluetooth System to record and submit their daily blood pressure and weight measurements to a mobile health nurse and research team. Subjects will be provided with the kit (Honeywell tablet, mobile hot spot, blood pressure cuff, and scale) at no cost. Subjects will participate in video telehealth visits at 48 hours and 7 days after discharge to help provide management for hypertension related issues.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive disorders of pregnancy including gestational, chronic, or preeclampsia diagnosed in the antenatal (primary admission for delivery of the baby (planned or due to hypertension) or postpartum period as determined by systolic blood pressure (SBP) greater than 140 or diastolic blood pressure (DBP) greater than 90 on two occasions 4 hours apart.
* Gestational age at time of delivery greater than 23 weeks gestation
* Postpartum with persistent SBP greater than 140 or DBP greater than 90 on two occasions 4 hours apart (to enroll would be prior to discharge from initial postpartum hospital stay).
* Primary hospital admission for the delivery of the neonate(s).

Exclusion Criteria:

* Inability to obtain informed consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 428 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Hoppe, DO, Principal Investigator — Clinical Assistant Professor
Locations (1):
- UnityPoint Health- Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoppe KK, Thomas N, Zernick M, Zella JB, Havighurst T, Kim K, Williams M, Niu B, Lohr A, Johnson HM. Telehealth with remote blood pressure monitoring compared with standard care for postpartum hypertension. Am J Obstet Gynecol. 2020 Oct;223(4):585-588. doi: 10.1016/j.ajog.2020.05.027. Epub 2020 May 19. No abstract available. PMID 32439388
- [Result] Thomas NA, Drewry A, Racine Passmore S, Assad N, Hoppe KK. Patient perceptions, opinions and satisfaction of telehealth with remote blood pressure monitoring postpartum. BMC Pregnancy Childbirth. 2021 Feb 19;21(1):153. doi: 10.1186/s12884-021-03632-9. PMID 33607957
- [Result] Hoppe KK, Williams M, Thomas N, Zella JB, Drewry A, Kim K, Havighurst T, Johnson HM. Telehealth with remote blood pressure monitoring for postpartum hypertension: A prospective single-cohort feasibility study. Pregnancy Hypertens. 2019 Jan;15:171-176. doi: 10.1016/j.preghy.2018.12.007. Epub 2018 Dec 31. PMID 30825917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2017 and July 2017, 55 women were enrolled into a feasibility study for the intervention (Aim 1). Through June 2018, a total of 428 women were enrolled in this study (214 in the intervention group including those from Aim 1 and 214 in the control group). Participants were recruited from Meriter Hospital in Madison, WI.
Groups:
- Mobile Health Participants: Participants used the mobile health device to record their blood pressure and weight measurements everyday for 6 weeks postpartum.
  Participants will have a video telehealth visit with the mobile health nurse at 48 hours and 7 days after discharge from the hospital.
Period: Aim 1: Feasibility and Satisfaction
Arm/Group | Mobile Health Participants | Standard of Care
Started | 55 | 0
Eligible Participants | 263 | 0
Participants Agreed to be Approached for Study | 124 | 0
Consented to Study | 55 | 0
Completed | 52 | 0
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0
Period: Aims 2-5: Intervention
Arm/Group | Mobile Health Participants | Standard of Care
Started (Aim 1 participants are included in the 214 participants enrolled and analyzed in Aims 2-5.) | 214 | 214
Number Analyzed | 214 | 214
Completed | 195 | 214
Not Completed | 19 | 0
Not completed — Withdrawal by Subject | 19 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mobile Health Participants: Participants will use the mobile health device to record their blood pressure and weight measurements everyday for 6 weeks postpartum.
  Participants will have a video telehealth visit with the mobile health nurse at 48 hours and 7 days after discharge from the hospital.
- Total: Total of all reporting groups
Arm/Group | Mobile Health Participants | Standard of Care | Total
Number analyzed (Participants) | 214 | 214 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.0) | 31.5 (5.5) | 31.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 214 | 428
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 202 | 199 | 401
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 10 | 12 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 25 | 41
  White | 175 | 168 | 343
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 214 | 214 | 428
Pre-pregnancy BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 31.8 [20.7 to 42.9] | 30.6 [20.2 to 41.0] | 31.2 [20.4 to 42.0]
Delivery BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 37.4 [24.2 to 50.6] | 36.6 [22.4 to 50.8] | 37.0 [23.3 to 50.7]
Primipara [Count of Participants; unit: Participants] — First time birth
  Participants | 108 | 91 | 199
Hypertension Classification [Count of Participants; unit: Participants]
  Chronic without Superimposed Preeclampsia | 21 | 23 | 44
  Chronic with Superimposed Preeclampsia | 22 | 23 | 45
  Gestational | 62 | 79 | 141
  Preeclampsia | 131 | 112 | 243
Other Subtypes of Hypertension of Interest [Count of Participants; unit: Participants]
  Mild Preeclampsia | 51 | 63 | 114
  Severe Preeclampsia | 80 | 49 | 129
  Hemolysis Elevated Liver enzyme Low Platelet (HELLP) | 11 | 1 | 12
  Eclampsia | 1 | 0 | 1
Married [Count of Participants; unit: Participants] | 163 | 149 | 312
Tobacco Use [Count of Participants; unit: Participants] | 12 | 21 | 33
Insurance Status [Count of Participants; unit: Participants]
  Private | 185 | 157 | 342
  Medicaid | 29 | 57 | 86
Pre-gestational Diabetes Mellitus [Count of Participants; unit: Participants] | 10 | 13 | 23
Gestational age at delivery [Count of Participants; unit: Participants]
  Preterm (less than 37 weeks) | 57 | 42 | 99
  Term (greater than or equal to 37 weeks) | 157 | 172 | 329

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Number of Participants Enrolled
Description: A goal of 55 participants enrolled into the mobile health program was set as a feasibility target.
Time Frame: up to 3 months
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Mobile Health Participants: Participants will use the mobile health device to record their blood pressure and weight measurements everyday for 6 weeks postpartum.
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 55

2. Primary Outcome: Aim 1: Number of Participants Who Completed the Study
Description: To assess retention, the number of participants who completed the study will be reported.
Time Frame: up to 6 weeks
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 52

3. Primary Outcome: Aims 2-5: Number of Participants Enrolled in 1 Year
Description: Aims 2-5 primary endpoint is enrollment of up to 40 participants at all times (for a total of 42 days) over one year (220 experimental and 220 matched controls for chart review).
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 214 | 214

4. Primary Outcome: Aims 2-5: Number of Participants With Hypertension-Related Hospital Readmissions
Description: Comparison of hypertension-related hospital readmissions between home telehealth with remote BP monitoring group and standard outpatient care during the first 6 weeks postpartum in women with hypertensive disorders of pregnancy (HDP).
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 1 | 8

5. Secondary Outcome: Aim 1: 6-week Hospital Readmission
Time Frame: up to 6 weeks
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 0

6. Secondary Outcome: Aim 1: Number of Participants With Severe Postpartum Hypertension After Discharge
Description: Defined using American College of Obstetricians and Gynecologists (ACOG) criteria blood pressure values of ≥160mmHg (systolic) or ≥110 mmHg (diastolic)
Time Frame: up to 6 weeks
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 9

7. Secondary Outcome: Aim 1: Number of Participants With Hypertension-Related Emergency Room Visits
Description: Comparison of hypertension-related emergency room visits between home telehealth with remote BP monitoring group and standard outpatient care during the first 6 weeks postpartum in women with HDP (hypertensive disorders of pregnancy).
Time Frame: up to 6 weeks postpartum
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 6

8. Secondary Outcome: Aim 1: Number of Participants With Need for Blood Pressure Treatment After Discharge
Description: Defined as participants having blood pressures exceeding the ACOG recommendations for blood pressure treatment (150/100 mmHg).
Time Frame: up to 6 weeks
Population: Aim 1 was an initial feasibility study enrolling 55 participants into the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 55
Participants | 29

9. Secondary Outcome: Aims 2-5: Number of Participants With Hypertension-Related Emergency Room Visits
Description: as for outcome 7
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 10 | 13

10. Secondary Outcome: Aims 2-5: Number of Participants With at Least One Blood Pressure Review Within 10 Days of Delivery
Description: Comparison of number of participants with at least one blood pressure review within 10 days of delivery between home telehealth with remote BP monitoring group and standard outpatient care during the first 6 weeks postpartum in women with HDP (hypertensive disorders of pregnancy).
Time Frame: up to 10 days of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 202 | 129

11. Secondary Outcome: Aims 2-5: Number of Participants on Antihypertensive Treatment Regimes
Description: Comparison of number of participants on antihypertensive treatments between home telehealth with remote BP monitoring group and standard outpatient care during the first 6 weeks postpartum in women with HDP (hypertensive disorders of pregnancy).
Time Frame: up to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 57 | 37

12. Secondary Outcome: Aims 2-5: Maximum Systolic Blood Pressure Intrapartum
Time Frame: Admission to delivery (up to 96 hours)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
mmHg | 160 [152 to 171] | 158 [151 to 167]

13. Secondary Outcome: Aims 2-5: Maximum Diastolic Blood Pressure Intrapartum
Time Frame: Admission to delivery (up to 96 hours)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
mmHg | 101 [96.0 to 110] | 102 [96.0 to 109]

14. Secondary Outcome: Aims 2-5: Systolic Blood Pressure at Discharge
Time Frame: Up to 96 hours postpartum
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
mmHg | 131 [124 to 138] | 129 [121 to 136]

15. Secondary Outcome: Aims 2-5: Diastolic Blood Pressure at Discharge
Time Frame: Up to 96 hours postpartum
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
mmHg | 78 [72 to 84] | 78 [71 to 84]

16. Secondary Outcome: Aims 2-5: Medication at Discharge
Time Frame: up to 96 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants
  Any Antihypertensive | 109 | 72
  Labetalol | 90 | 61
  Nifedipine | 39 | 20

17. Secondary Outcome: Aims 2-5: Postpartum Day of Discharge
Time Frame: up to 4.5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
days | 3.35 (1.2) | 2.92 (1.1)

18. Secondary Outcome: Aims 2-5: Inpatient Nonsteroidal Anti-inflammatory Drug (NSAID) Use
Time Frame: up to 4 days post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 186 | 189

19. Secondary Outcome: Aims 2-5: Change in Weight From First Prenatal Care Visit to Delivery
Time Frame: first prenatal care visit (on average 8-14 weeks of pregnancy, delivery (on average 37-40 weeks of pregnancy)
Population: Number of participants for which both first prenatal care weight and delivery weight were measured.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 212 | 210
kilograms | 14.6 (8.0) | 14.4 (8.4)

20. Secondary Outcome: Self-Administered Questionnaire Satisfaction Survey Scores
Description: In collaboration with the University of Wisconsin Survey Center, the investigators developed a 37-question self-administered questionnaire (SAQ) satisfaction survey to all participants at the 6-week postpartum clinic visit. The survey utilized a variety of question formats including Likert scales with response ranging from 1 to 5 ("Not at all"; "A little"; "Somewhat"; "Quite a bit"; "A great deal" or "Never"; "Rarely"; "Sometimes"; "Very often"; "Extremely often"), dichotomous questions with a Yes/No response, and free text. A summary of mean scores (1-5) are reported here.
Time Frame: up to 6 weeks postpartum
Population: Of the 214 participants enrolled in the intervention, 128 participants responded to the 6 week postpartum survey. Not all questions were answered by all survey respondents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 128
score on a scale
  How complicated are mHealth's instructions?: number analyzed (Participants) | 127
  How complicated are mHealth's instructions? | 0.25 (0.67)
  How much mental effort does mHealth require?: number analyzed (Participants) | 127
  How much mental effort does mHealth require? | 0.59 (0.74)
  How easily does mHealth fit into your lifestyle?: number analyzed (Participants) | 127
  How easily does mHealth fit into your lifestyle? | 2.65 (0.96)
  How easy was it to get help?: number analyzed (Participants) | 43
  How easy was it to get help? | 3.33 (0.87)
  How confident do you feel using the mHealth devices?: number analyzed (Participants) | 127
  How confident do you feel using the mHealth devices? | 3.46 (0.79)
  How hard is the monitor to use?: number analyzed (Participants) | 126
  How hard is the monitor to use? | 0.16 (0.49)
  How organized is the monitor?: number analyzed (Participants) | 127
  How organized is the monitor? | 3.27 (0.78)
  How helpful are the monitor's prompts?: number analyzed (Participants) | 127
  How helpful are the monitor's prompts? | 2.57 (1.34)
  How easy is the blood pressure cuff to use?: number analyzed (Participants) | 127
  How easy is the blood pressure cuff to use? | 3.44 (0.79)
  How hard is the weight scale to use?: number analyzed (Participants) | 126
  How hard is the weight scale to use? | 0.37 (1.06)
  How reasonable is the amount of time it takes to record your blood pressure?: number analyzed (Participants) | 127
  How reasonable is the amount of time it takes to record your blood pressure? | 3.46 (0.77)
  How reasonable is the amount of time it takes to record your weight?: number analyzed (Participants) | 127
  How reasonable is the amount of time it takes to record your weight? | 3.47 (0.79)
  How burdensome is it to record your blood pressure daily?: number analyzed (Participants) | 127
  How burdensome is it to record your blood pressure daily? | 0.85 (0.93)
  How burdensome is it to record your weight daily?: number analyzed (Participants) | 127
  How burdensome is it to record your weight daily? | 0.78 (0.98)
  How secure do you feel submitting your vitals?: number analyzed (Participants) | 127
  How secure do you feel submitting your vitals? | 3.41 (0.76)
  How much more in control of your own health do you feel? | 2.91 (0.9)
  How much more aware of your own health do you feel? | 3.30 (0.74)
  Do you prefer going to clinic/hospital instead of using mHealth for postpartum follow-up? | 0.31 (0.78)
  How much would you recommend mHealth to others in your situation?: number analyzed (Participants) | 127
  How much would you recommend mHealth to others in your situation? | 3.49 (0.79)
  How enjoyable are the mHealth devices to use?: number analyzed (Participants) | 127
  How enjoyable are the mHealth devices to use? | 2.41 (1.06)
  How satisfied are you with the mHealth devices?: number analyzed (Participants) | 127
  How satisfied are you with the mHealth devices? | 3.32 (0.83)
  To what extent does using the mHealth tech make you feel safer? | 2.86 (0.96)
  How often do you feel unsafe while using mHealth?: number analyzed (Participants) | 8
  How often do you feel unsafe while using mHealth? | 0.38 (1.06)
  How fun is answering questions using the Genesis Touch Monitor?: number analyzed (Participants) | 127
  How fun is answering questions using the Genesis Touch Monitor? | 2.24 (1.03)
  Did the Genesis Touch Monitor have all functions you expected?: number analyzed (Participants) | 127
  Did the Genesis Touch Monitor have all functions you expected? | 3.02 (0.98)
  Do you like the touch screen technology on the Genesis Touch monitor?: number analyzed (Participants) | 127
  Do you like the touch screen technology on the Genesis Touch monitor? | 3.43 (0.74)
  Does using mHealth make you worry more, less or the same? | 1.23 (0.63)

21. Secondary Outcome: Participant Counts for Relevant SAQ Satisfaction Survey Questions
Description: In collaboration with the University of Wisconsin Survey Center, the investigators developed a 37-question self-administered questionnaire (SAQ) satisfaction survey to all participants at the 6-week postpartum clinic visit. The survey utilized a variety of question formats including Likert scales with response ranging from 1 to 5 ("Not at all"; "A little"; "Somewhat"; "Quite a bit"; "A great deal" or "Never"; "Rarely"; "Sometimes"; "Very often"; "Extremely often"), dichotomous questions with a Yes/No response, and free text. A summary of questions with participant counts is reported here.
Time Frame: up to 6 weeks postpartum
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants
Number analyzed (Participants) | 128
Participants
  Number of Participants who got help for problems with their devices: number analyzed (Participants) | 67
  Number of Participants who got help for problems with their devices | 24
  Number of Participants for whom it took 1 minute to measure their blood pressure | 118
  Number of Participants for whom it took 5 minutes to measure their blood pressure | 11
  Number of Participants for whom it took 1 minute to measure their weight | 122
  Number of Participants for whom it took 5 minutes to measure their weight | 5
  Number of Participant who had any problems using the Genesis Touch monitor: number analyzed (Participants) | 127
  Number of Participant who had any problems using the Genesis Touch monitor | 49
  Number of Participants who had any problems using the blood pressure cuff: number analyzed (Participants) | 127
  Number of Participants who had any problems using the blood pressure cuff | 108
  Number of Participants who had any problems using the scale: number analyzed (Participants) | 127
  Number of Participants who had any problems using the scale | 107
  Number of Participants who had concerns sending their vitals to their health care provider: number analyzed (Participants) | 127
  Number of Participants who had concerns sending their vitals to their health care provider | 4
  Number of Participants who had enough control over their data | 113
  Number of Participant who had to go to an emergency room after discharge | 14
  Number of Participants who had a hospital readmission | 3
  Number of Participants who went to a different hospital than their delivery hospital: number analyzed (Participants) | 3
  Number of Participants who went to a different hospital than their delivery hospital | 1

22. Other Pre Specified Outcome: Cost Effective Analysis on Remote Patient Monitoring for Postpartum Hypertension.
Description: Cost effectiveness modeling will be performed to determine whether it is cost effective to use remote patient modeling for women with postpartum hypertension in comparison to standard outpatient care in women with hypertension-related disorders of pregnancy.
Time Frame: Up to 12 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Mode of Delivery
Time Frame: at delivery (on average 37-40 weeks of pregnancy)
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants
  Vaginal spontaneous | 84 | 112
  Cesarean | 114 | 87
  Operative vaginal | 16 | 15

24. Other Pre Specified Outcome: Neonatal Birthweight
Time Frame: at time of birth
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
grams | 3180 [2660 to 3540] | 3060 [2610 to 3490]

25. Other Pre Specified Outcome: Neonatal Intensive Care Unit Admissions
Time Frame: at birth
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Participants | Standard of Care
Number analyzed (Participants) | 214 | 214
Participants | 67 | 55

ADVERSE EVENTS:
Time Frame: up to 6 weeks post partum
Arm/Group | Mobile Health Participants | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/214
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/214
Other Adverse Events (participants affected / at risk) | 0/214 | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03111095/Prot_SAP_000.pdf